CLINICAL TRIAL: NCT06885892
Title: Posterior Tibial Artery Perforator-Pedicled Propeller Flaps for Reconstruction of the Defects in the Lower Leg（Case Series）
Brief Title: Posterior Tibial Artery Perforator-Pedicled Propeller Flaps in Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2015-JS018-01
Record Dates: First submitted 2025-03-09; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Trauma Patients with Soft Tissue Defects
Keywords: the lower leg; soft tissue defects; perforator flaps; propeller flaps; doppler ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- surgery (Experimental): posterior tibial artery perforator-pedicled propeller flaps transplantation for soft-tissue defects
  Interventions: Procedure: Posterior Tibial Artery Perforator-Pedicled Propeller Flaps; Procedure: Perforator-Pedicled Propeller Flaps

INTERVENTIONS:
Procedure: Posterior Tibial Artery Perforator-Pedicled Propeller Flaps — Posterior tibial artery perforator-pedicled propeller flaps are feasible, safe, and effective procedure in the reconstruction of the defects in the lower leg.
Procedure: Perforator-Pedicled Propeller Flaps — Posterior Tibial Artery Perforator-Pedicled Propeller Flaps

SUMMARY:
Soft tissue defects in the lower leg remain a challenge for surgeons due to frequent bone exposure and paucity of soft tissues. The goal in this study was to evaluate the surgical technique and clinical significance of posterior tibial artery perforator-pedicled propeller flaps for reconstruction of defects in the lower leg.

DETAILED DESCRIPTION:
The construction of the lower extremity defects with exposed bone and tendon is considered as the biggest challenge of all body regions in many plastic and reconstructive surgeons. The lower leg regions are in visible areas. Defects recovery and aesthetic consideration should be considered at the same time with the development of the economy and society. Although free flaps have been used to reconstruct these defects, some disadvantages still exist, such as needing microinstruments, long operation time and none like-with-like repair. In this article, a series of patients with soft tissue defects in the lower leg were transplanted with posterior tibial artery perforator-pedicled propeller flaps.

ELIGIBILITY:
Inclusion Criteria:

* 1.age range :10-80years. 2. in good overall heath without severe comorbidities. 3. posterior perforator tibial artery is no damage.

Exclusion Criteria:

1. age range <10years or >80years.
2. with severe comorbidities
3. Posterior perforator tibial artery of panticipants is damage

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
flaps observation | 12-24months
  flaps color :normal;pale;cyanoderma

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin J, Zhou F, Sun YD, Gao YS, Li HZ, Zheng HP, Zhang YF, Li QF, Ward PJ, Yang YL, Liu CY. Modified Anterior Tibial Artery Perforator-Pedicled Propeller Flap for Soft-Tissue Coverage of the Ankle and Heel. World J Surg. 2020 Jul;44(7):2237-2242. doi: 10.1007/s00268-020-05452-y. PMID 32123981
- [Background] Jakubietz RG, Jakubietz MG, Gruenert JG, Kloss DF. The 180-degree perforator-based propeller flap for soft tissue coverage of the distal, lower extremity: a new method to achieve reliable coverage of the distal lower extremity with a local, fasciocutaneous perforator flap. Ann Plast Surg. 2007 Dec;59(6):667-71. doi: 10.1097/SAP.0b013e31803c9b66. PMID 18046150